CLINICAL TRIAL: NCT04325334
Title: Linking Biomechanical and Imaging Outcomes to Better Understand the Effects of Running on Knee Joint Health
Brief Title: Osteoarthritis Running & Cartilage Assessment
Acronym: ORCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Hunt, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-01806
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; running; magnetic resonance imaging; MRI
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Both runners with and without knee osteoarthritis will be recruited. They will all receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Running volume increase (Experimental): Participants will be be given a running program based on their running mileage on inclusion and supported by regular contacts with the study trainer.
  Interventions: Behavioral: Running volume increase

INTERVENTIONS:
Behavioral: Running volume increase — Participants will receive a 12-week running program to increase their running volume by approximately 10% per week on average, and in accordance with the "10% rule" advocated to minimize injury rates. For the purpose of this study, participants will run using their habitual technique - i.e. no specific instructions on 'how' to run will be provided; rather, they will simply be instructed on 'how much' to run.

SUMMARY:
Knee osteoarthritis (OA) is a debilitating disease affecting millions of Canadians. Exercise is a core treatment for knee OA, and is advocated by all clinical guidelines. However, the safety of recreational running in the presence of knee OA is unclear. There are no studies available to provide direct data to appropriately inform runners and clinicians whether running should be advocated for joint health. Our research study will address this gap.

ELIGIBILITY:
Inclusion Criteria:

ALL:

* aged greater than 40 years
* recreational runners who run at least twice per week for a total of at least 10 km, and have done so for a minimum of 12 months
* comfortable running on a treadmill for 30 minutes.

TFOA Group:

* exhibit radiographic evidence of mild or moderate tibiofemoral osteoarthritis (TFOA) according to the Kellgren and Lawrence OA classification scale (grade ≥ 2)
* report knee pain on most days of the previous 3 months (during running and activities of daily living).

Control Group:

* free of any radiographic signs of TFOA according to the Kellgren and Lawrence scale (grade = 0)
* pain free in both knees for the 12 months prior to recruitment.

Exclusion Criteria:

ALL:

* any history of traumatic knee injury (fracture, severe sprain, meniscus injury)
* presence of an inflammatory arthritic condition
* presence of any health condition (other than OA in the TFOA group) affecting normal movement or precludes engaging in moderate to high impact activities such as running
* use of any oral or injected corticosteroids or viscosupplementation in the previous 6 months
* any history of surgery in either knee
* standard contra-indications to magnetic resonance imaging (MRI).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 12 weeks in T2 relaxation time of the medial femoral cartilage | Baseline, 12 weeks
  T2 relaxation represents the time constant of the molecular motion of water in cartilage, which is influenced by the composition of collagen and specifically reflects changes to the extracellular matrix. This constant is assessed using MRI.
Change from Baseline to 12 weeks in T2 relaxation time of the medial tibial cartilage | Baseline, 12 weeks
  T2 relaxation represents the time constant of the molecular motion of water in cartilage, which is influenced by the composition of collagen and specifically reflects changes to the extracellular matrix. This constant is assessed using MRI.
Change from Baseline to 12 weeks in T2 relaxation time of the lateral femoral cartilage | Baseline, 12 weeks
  T2 relaxation represents the time constant of the molecular motion of water in cartilage, which is influenced by the composition of collagen and specifically reflects changes to the extracellular matrix. This constant is assessed using MRI.
Change from Baseline to 12 weeks in T2 relaxation time of the lateral tibial cartilage | Baseline, 12 weeks
  T2 relaxation represents the time constant of the molecular motion of water in cartilage, which is influenced by the composition of collagen and specifically reflects changes to the extracellular matrix. This constant is assessed using MRI.

SECONDARY OUTCOMES:
Change from Baseline to 12 weeks in T1ρ relaxation time of the medial femoral cartilage | Baseline, 12 weeks
  T1ρ provides an indication of glycosaminoglycan concentration in cartilage assessed using MRI.
Change from Baseline to 12 weeks in T1ρ relaxation time of the medial tibial cartilage | Baseline, 12 weeks
  T1ρ provides an indication of glycosaminoglycan concentration in cartilage assessed using MRI.
Change from Baseline to 12 weeks in T1ρ relaxation time of the lateral femoral cartilage | Baseline, 12 weeks
  T1ρ provides an indication of glycosaminoglycan concentration in cartilage assessed using MRI.
Change from Baseline to 12 weeks in T1ρ relaxation time of the lateral tibial cartilage | Baseline, 12 weeks
  T1ρ provides an indication of glycosaminoglycan concentration in cartilage assessed using MRI.
Change from Baseline to 12 weeks in knee joint loading: peak knee adduction moment | Baseline, 12 weeks
  Participants will run on an instrumented treadmill in their habitual running shoes while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and treadmill-embedded force platforms.
Change from Baseline to 12 weeks in knee joint loading: knee adduction moment impulse | Baseline, 12 weeks
  Participants will run on an instrumented treadmill in their habitual running shoes while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and treadmill-embedded force platforms.
Change from Baseline to 12 weeks in knee joint loading: peak flexion moment | Baseline, 12 weeks
  Participants will run on an instrumented treadmill in their habitual running shoes while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and treadmill-embedded force platforms.
Change from Baseline to 12 weeks in knee joint loading: flexion moment impulse | Baseline, 12 weeks
  Participants will run on an instrumented treadmill in their habitual running shoes while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and treadmill-embedded force platforms.
Change from Baseline to 12 weeks in knee joint kinematics: peak knee flexion angle | Baseline, 12 weeks
  Participants will run on an instrumented treadmill in their habitual running shoes while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and treadmill-embedded force platforms.
Change from Baseline to 12 weeks in knee joint kinematics: knee joint angle excursion | Baseline, 12 weeks
  Participants will run on an instrumented treadmill in their habitual running shoes while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and treadmill-embedded force platforms.
Change from Baseline to 12 weeks in foot strike pattern | Baseline, 12 weeks
  Participants will run on an instrumented treadmill in their habitual running shoes while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and treadmill-embedded force platforms.
Change from Baseline to 12 weeks in step rate | Baseline, 12 weeks
  Participants will run on an instrumented treadmill in their habitual running shoes while analyzed using three-dimensional motion analysis. Kinematic (joint angle) and kinetic (joint loading) data will be collected synchronously using high-speed digital cameras and treadmill-embedded force platforms.
Change from Baseline to 12 weeks in knee symptoms: Knee Osteoarthritis Outcome Score (KOOS) | Baseline, 12 weeks
  Validated questionnaire on symptoms and functional limitations related to knee osteoarthritis. The score is expressed in percentage (0-100), with 0 representing extreme knee problems and 100 representing no knee problems.
Change from Baseline to 12 weeks in knee symptoms: Visual Analog Scale | Baseline to 12 weeks, averaged weekly
  Knee pain during and after running will be assessed for each training. The minimum value is "No Pain" and the maximum value is "Worst Pain Imaginable". Each week of training will be averaged.
Change from Baseline to 12 weeks in weekly running distance | Baseline to 12 weeks, averaged weekly
  Participants will record their weekly running distance using an online diary.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Hunt, PT, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Motion Analysis and Biofeedback Laboratory, The University of British Columbia, Vancouver, British Columbia, Canada

DOCUMENTS (2):
  • Study Protocol (2019-11-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT04325334/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT04325334/SAP_001.pdf